CLINICAL TRIAL: NCT00828334
Title: Transcatheter Occlusion of Patent Ductus Arteriosus (PDA) With the NIT-OCCLUD PDA Occlusions System
Brief Title: NIT-OCCLUD PDA Phase II Sentinel Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PFM Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G010278
Record Dates: First submitted 2009-01-20; First posted 2009-01-23 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Ductus Arteriosus, Patent
Keywords: transcatheter occlusion of patent ductus arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcatheter PDA Coil (Experimental): Transcatheter occlusion of Patent Ductus Arteriosus (PDA) with the flex and medium Nit-Occlud PDA.
  Interventions: Device: Transcatheter PDA Coil

INTERVENTIONS:
Device: Transcatheter PDA Coil — The Nit-Occlud PDA is a permanently implanted prosthesis indicated for percutaneous, transcatheter closure of small to moderate size patent ductus arteriosus with a minimum angiographic diameter < 4 mm.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Nit-Occlud -PDA Occlusion System for transcatheter closure of PDA with minimum angiographic diameter less than 4 mm, and to compare one year safety and efficacy outcomes with recommended OPCs.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate whether transcatheter occlusion of PDAs with a minimum vessel diameter of 4 mm or smaller, by means of permanent implantation of the Nit-Occlud Spiral Coil for PDA Occlusion, is safe and effective.

The device used for this purpose is a set of two items named "Nit-Occlud - PDA Occlusion System":

* Nit-Occlud coils, 2 types: flexible (3 sizes) and medium (3 sizes)
* Introducer Sheath, F4 or F5 85cm.

The intended use of the device is the percutaneous, transluminal closure of PDA with an internal diameter or 4mm and smaller in patients who comply with the selection criteria.

The investigation will continue until the sponsor receives FDA approval for commercial distribution and implantation of the system, or until the project is terminated by the sponsor or by the investigators.

The objectives of this study are:

1. To determine the safety of the spiral coil by monitoring and reporting deaths and adverse events associated with the device and device placement.
2. To determine the effectiveness of the spiral coil by evaluating clinical and echocardiographic occlusion rates.

ELIGIBILITY:
Inclusion Criteria:

* PDA with 4 mm or smaller minimum diameter by color Doppler
* Patent weight > 5 Kg, Age 6 months to 21 years (Patients older than 21 years may have device implant and be included in a study registry.)
* Previous treatment by surgery or Nit-Occlud device with residual PDA noted at least 6 months after the procedure
* Angiographic minimum PDA diameter (D1) less than 4 mm. (Patients with angiographic diameters larger than 4 mm and smaller or equal to 5 mm may have device implant and be included in a study registry.)

Exclusion Criteria:

* Associated cardiac anomalies requiring surgery
* Known bleeding or blood clotting disorders
* Ongoing febrile illness
* Pregnancy
* Pulmonary hypertension/increased pulmonary vascular resistance (>5 Wood Units)
* Known hypersensitivity to contrast medium

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 357 (Actual)
Dates: Start 2002-11; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Objective Performance Criteria (OPC) Technical Success at Implant | One year
Clinical Closure and Echocardiographic Closure at 12 month follow-up | One year
Serious Adverse Events and Mortality at 12 months | One year
Total Device or Procedure Related Adverse Events | One year

SECONDARY OUTCOMES:
Composite Success. That is technical success, clinical and echocardiographic closure, and absence of device or procedure related death or serious AE at 12 months follow-up | One year

CONTACTS AND LOCATIONS:
Overall Officials: John W Moore, MD, MPH, Principal Investigator — Rady Children's Hospital, San Diego, Department of Pediatrics, UCSD, School of Medicine
Locations (15):
- United States (15):
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - A.I. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Children's Hospital of Illinois, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital of Iowa, Iowa City, Iowa
  - Children's Hospital of Akron, Akron, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Children's Medical Center of Dallas, Dallas, Texas
  - Children's Hospital and Regional Medical Center Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided